CLINICAL TRIAL: NCT07246850
Title: A Randomized, Triple-blind, Placebo-controlled Study to Evaluate the Effects of a Throat Spray on the Incidence and Duration of Sickness
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beekeeper's Naturals Inc (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20694
Record Dates: First submitted 2025-11-19; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Sore-throat; Common Cold
MeSH Terms: conditions — Pharyngitis; Common Cold

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beekeeper's Propolis Throat Spray (Experimental)
  Interventions: Dietary Supplement: Beekeeper's Propolis Throat Spray
- Placebo Throat Spray (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo Throat Spray

INTERVENTIONS:
Dietary Supplement: Beekeeper's Propolis Throat Spray — Participants will administer four sprays of Beekeeper's Propolis Throat Spray into the back of the mouth once daily in the morning for 16 weeks.
  Arms: Beekeeper's Propolis Throat Spray
Dietary Supplement: Placebo Throat Spray — Participants will administer four sprays of a placebo throat spray into the back of the mouth once daily in the morning for 16 weeks.
  Arms: Placebo Throat Spray

SUMMARY:
This is a randomized, triple-blind, placebo-controlled clinical trial evaluating the effects of Beekeeper's Naturals Propolis Immune Support Throat Spray on the incidence and duration of sickness over a 16-week period. The study will enroll 100 healthy adults aged 18 to 65.

ELIGIBILITY:
Inclusion Criteria:

* Be male or female
* Be aged 18-65
* Meet at least one of the following criteria:

Work in a hospital or other healthcare setting Work in a school

* Have a child/children under the age of 10
* Be willing to take the test or placebo product once daily and complete study questionnaires every four weeks for the 16-week study period
* Be willing to refrain from taking any over-the-counter products, herbal remedies, or supplements that target immune function during the study period and for two weeks prior.
* Be willing to maintain their current diet, sleep schedule, and activity level for the duration of the study.
* Be in good general health and not live with any uncontrolled chronic conditions.
* Reside in the United States.

Exclusion Criteria:

* Has undergone any surgeries or invasive treatments in the past six months or plans to undergo any during the study period
* Anyone with seasonal allergies
* Anyone who follows a restrictive diet (e.g., keto, vegan, raw, carnivore, etc.).
* Anyone who got a vaccination in the last 2 weeks.
* Anyone taking one or more prescription medications:

Corticosteroids: Prednisone (prednisone), Deltasone (prednisolone), Medrol (methylprednisolone), Decadron (dexamethasone), Cortef (hydrocortisone), Kenalog (triamcinolone), Flonase (fluticasone), Nasonex (mometasone) Biologics (Immunomodulating Agents): Humira (adalimumab), Enbrel (etanercept), Remicade (infliximab), Stelara (ustekinumab), Cosentyx (secukinumab), Taltz (ixekizumab), Orencia (abatacept), Simponi (golimumab), Xeljanz (tofacitinib), Rituxan (rituximab), Actemra (tocilizumab), Kineret (anakinra) DMARDs (Disease-Modifying Antirheumatic Drugs): Methotrexate (methotrexate), Plaquenil (hydroxychloroquine), Arava (leflunomide), Azulfidine (sulfasalazine), Imuran (azathioprine), CellCept (mycophenolate mofetil), Cytoxan (cyclophosphamide) JAK Inhibitors: Olumiant (baricitinib), Rinvoq (upadacitinib), Jakafi (ruxolitinib) Other Immunosuppressive Medications: Prograf (tacrolimus), Neoral, Sandimmune (cyclosporine), Rapamune (sirolimus), Zortress (everolimus)

* Has had any major illness in the past three months.
* Drinks heavily (defined as 8 or more alcoholic drinks per week for women or 15 or more alcoholic drinks per week for men).
* Uses illicit drugs.
* Has known allergies or hypersensitivities to any of the study product ingredients.
* Is immunocompromised due to a medical condition or due to immunosuppressive medications or treatments.
* Has any known autoimmune conditions.
* Has any chronic health conditions that could impact participation in the study, including cancer, liver, or mental health disorders.
* Has known serious allergic reactions requiring the use of an Epi-Pen.
* Is currently pregnant, trying to conceive, or breastfeeding.
* Is currently participating in another research study or plans to do so during the 16-week study period.
* Has a history of substance abuse.
* Is currently a smoker or has been a smoker in the past three months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-12-30 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Changes in incidence and duration of sickness | Baseline, Weeks 4, 8, 12, and 16
  Self-reported via questionnaires comparing frequency and duration of illness episodes between groups

SECONDARY OUTCOMES:
Perceived improvement in overall health | Baseline, Week 4, Week 8, Week 12, and Week 16
  Participants will report perceived changes in their overall health using self-administered questionnaires.
Perceived improvement in overall well-being | Baseline, Week 4, Week 8, Week 12, and Week 16
  Participants will report their sense of overall well-being using self-administered questionnaires throughout the study.
Perceived immune system support | Baseline, Week 4, Week 8, Week 12, and Week 16
  Participants will rate their perception of immune system support using self-administered questionnaires during the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Las Vegas, Nevada, United States